CLINICAL TRIAL: NCT00867295
Title: A Randomized, Double-blind, Placebo-controlled Trial to Determine Effectiveness of Antibiotic Prophylaxis for Totally Implantable Venous Access Device.
Brief Title: Effectiveness of Antibiotic Prophylaxis for Totally Implantable Venous Access Device
Acronym: TIVAD
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Istanbul University (Other)
Responsible Party: Istanbul University Institute of Oncology (Hasan Karanlik, MD), Istanbul University Institute of Oncology
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2009/22
Record Dates: First submitted 2009-03-20; First posted 2009-03-23 (Estimated); Last update posted 2010-06-02 (Estimated); Status verified 2009-03

CONDITIONS: Solid Tumor
Keywords: implantable catheters; Indwelling Catheters; infection; cefazolin sodium; prophylactic; antibiotic; totally implantable venous access device; cancer patients
MeSH Terms: conditions — Infections | interventions — Cefazolin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- placebo (Placebo Comparator): no antibiotic is used
  Interventions: Drug: placebo
- drug (Active Comparator): cefazolin Sodium 1g i.v. before the operation
  Interventions: Drug: cefazolin Sodium

INTERVENTIONS:
Drug: cefazolin Sodium — cefazolin Sodium 1g i.v. before operation
  Arms: drug
Drug: placebo — placebo
  Arms: placebo

SUMMARY:
This randomized trial is determining the role of antibiotic prophylaxis in the prevention of the infectious complications in patients carrying out totally implantable venous access device.

ELIGIBILITY:
Inclusion Criteria:

* Older than 18 years of age
* Have solid tumor
* White cells >4000
* Platelets >100.000
* Prothrombin time in normal range

Exclusion Criteria:

* Drug allergy
* Diabetes mellitus

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2008-09; Primary Completion 2009-12 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
infectious complication | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Hasan Karanlik, MD, Principal Investigator — Istanbul University Institute of Oncology Department of Surgery
Locations (1):
- Istanbul University Institute of Oncology, Istanbul, Capa, Turkey (Türkiye)

REFERENCES:
- [Derived] Karanlik H, Kurul S, Saip P, Unal ES, Sen F, Disci R, Topuz E. The role of antibiotic prophylaxis in totally implantable venous access device placement: results of a single-center prospective randomized trial. Am J Surg. 2011 Jul;202(1):10-5. doi: 10.1016/j.amjsurg.2010.05.005. Epub 2011 May 23. PMID 21601826